CLINICAL TRIAL: NCT06773247
Title: Effectiveness of Myofascial Release Technique Versus Dry Cupping Therapy in Management of Patients with Non-Specific Low Back Pain
Brief Title: Effectiveness of Myofascial Release Versus Dry Cupping in Management of Non-Specific Low Back Pain
Acronym: NSLBP-MFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rabab Ali Mohamed, Assistant Professor of Physical Therapy, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (P.T. REC/012/005495)
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Non-specific Low Back Pain
Keywords: Myofascial Release, Cupping, NSLBP

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Myofascial Release Technique (Experimental): Vertical stroking technique was performed in lumbar region to quadratus lumborum. Activities like sustained repetitive movements, twisting, bending, sedentary posture for prolonged duration, muscle imbalance, etc. leads to trigger point formation making quadratus lumborum as a common source of low back pain. It was performed as follow; Quadratus lumborum is palpated in prone and side lying for trigger points. The technique is applied by the patient positioned in side lying with a pillow under waist to exaggerate stretch of the muscle.
  Interventions: Other: I. Myofascial Release Technique ,Cupping Technique and II. Conventional Physical Therapy

INTERVENTIONS:
Other: I. Myofascial Release Technique ,Cupping Technique and II. Conventional Physical Therapy — The cupping procedure was performed as follows: Massage oil was applied over the area first to improve contact and makes it easier to move the cup's position. double-walled glass cups (6 glasses with diameters from 75 to 100 mm) were held inverted, after which each glass was placed on an afflicted area overlying the low back muscle (acupoint: BL23).
  Myofascial Release Technique Vertical stroking technique was performed in lumbar region to quadratus lumborum. AIt was performed as follow; Quadratus lumborum is palpated in prone and side lying for trigger points. The technique is applied by the patient positioned in side lying with a pillow under waist to exaggerate stretch of the muscle. The therapist stands at level of patient's hip posterior and counter pre

SUMMARY:
Objective: The aim of this study was to compare the differences between the effect of myofascial release technique versus cupping technique on pain intensity level, spinal mobility and functional disabilities level in patients with NSLBP.

Methods: The study participants were 60 patients from both genders diagnosed as NSLBP. Their age ranged from 45 to 55 years old. They were assigned randomly into two groups: Group A (MFR): 20 patients received MFR and conventional physical therapy treatment. Group B: 20 patients received cupping technique and conventional physical therapy treatment. Group C: 20 patients received conventional physical therapy treatment only. All groups received treatment protocols three times a week for 4 consecutive weeks.

DETAILED DESCRIPTION:
The study participants were assigned randomly into two groups; Group A: 20 patients received MFR and conventional physical therapy treatment (therapeutic exercises in the form of stretching exercises for the back, iliopsoas, and hamstring muscles and strengthening exercises for the abdominal muscles for 30 minutes. Group B: 20 patients received cupping technique and conventional physical therapy treatment (therapeutic exercises in form of stretching exercises for the back, iliopsoas, and hamstring muscles and strengthening exercises for the abdominal muscles for 30 minutes. Group C: 20 patients received conventional physical therapy treatment only (therapeutic exercises in form of stretching exercises for the back, iliopsoas, and hamstring muscles and strengthening exercises for the abdominal muscles for 30 minutes. All groups received treatment protocols three times a week for 4 consecutive weeks.

Intervention I. Myofascial Release Technique Vertical stroking technique was performed in lumbar region to quadratus lumborum. Activities like sustained repetitive movements, twisting, bending, sedentary posture for prolonged duration, muscle imbalance, etc. leads to trigger point formation making quadratus lumborum as a common source of low back pain. It was performed as follow; Quadratus lumborum is palpated in prone and side lying for trigger points. The technique is applied by the patient positioned in side lying with a pillow under waist to exaggerate stretch of the muscle. The therapist stands at level of patient's hip posterior and counter pressure was applied by one hand on the ribs in a cephalic direction and with the other hand vertical stroking was performed by the knuckles caudally through its course in direction of the barrier. When a barrier was reached, light pressure was maintained to stretch the barrier and wait for approximately 3-5 minutes. Prior to release, a therapeutic pulse was felt (e.g. heat). As the barrier releases, the hand felt the motion and softening of the tissue. Sessions were conducted three days / week every other day for four weeks Cupping Technique The cupping procedure was performed as follows: Massage oil was applied over the area first to improve contact and makes it easier to move the cup's position. double-walled glass cups (6 glasses with diameters from 75 to 100 mm) were held inverted, after which each glass was placed on an afflicted area overlying the low back muscle (acupoint: BL23. This point is located 1.5 cm lateral to the posterior midline, on the level of the lower border of the spinous process of the second lumbar vertebra) and has been used to treat conditions such as lower back pain. As the air inside the cups cooled, vacuums were created, drawing up the skin within each cup. The cups were separated by 1-2 centimeters. The glasses were removed after 10 to 20 minutes depending on the colour of the circular so-called cupping marks, which range from slightly rose to dark pink. During cupping, the patients were asked to remain as still as possible. If the suctioning became too painful to bear, the cups were removed before the full time had elapsed.

II. Conventional Physical Therapy Treatment It consists of stretching exercises for the back, iliopsoas, and hamstring muscles and strengthening exercises for the abdominal muscles for 30 minutes. Three sets of stretching exercises, each involving a 30-sec hold and 30 sec of rest repeated three times, were performed in three sessions per week over four weeks. One set of strengthening exercises, consisting of 10 repetitions with a 5-sec hold, sessions were conducted three days a week, every other day, for four weeks.

The cupping procedure was performed as follows: Massage oil was applied over the area first to improve contact and makes it easier to move the cup's position. double-walled glass cups (6 glasses with diameters from 75 to 100 mm) were held inverted, after which each glass was placed on an afflicted area overlying the low back muscle (acupoint: BL23. This point is located 1.5 cm lateral to the posterior midline, on the level of the lower border of the spinous process of the second lumbar vertebra) and has been used to treat conditions such as lower back pain. As the air inside the cups cooled, vacuums were created, drawing up the skin within each cup. The cups were separated by 1-2 centimeters. The glasses were removed after 10 to 20 minutes depending on the colour of the circular so-called cupping marks, which range from slightly rose to dark pink. During cupping, the patients were asked to remain as still as possible. If the suctioning became too painful to bear, the cups were removed before the full time has elapsed. Cupping therapy was performed for 15-20 minutes three days / week every other day for four weeks

ELIGIBILITY:
Inclusion criteria:

1. patients age ranged from 45 to 55 years old and body mass index of 18.5-24.9 (kg/m2) with NSLBP of 3 or more month's duration.
2. All patients reported pain score of 4-6 based on the visual analog scale (VAS). 3.Patient with limitation in range of motion of lumbar spine due to tightness of the muscles, hypersensitive tender points on palpation along with pain localized para spinally .

Exclusion criteria:

1. Patients presented with lumbar radiculopathy
2. spinal pathology (fracture or tumors) or history of any spinal surgery
3. lumbar canal stenosis, osteoporosis
4. pregnancy related back pain, and spinal deformities like scoliosis or kyphosis.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-03 (Estimated); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-04-03 (Estimated)

PRIMARY OUTCOMES:
pain in low back area | 4 weeks
  Visual analog scale (VAS) was used to assess the intensity of perceived pain pre and post treatment in patients with NSLBP. The VAS is a reliable and valid tool for the quantification of perceived pain

SECONDARY OUTCOMES:
Functional Disability | 4 weeks
  Level of daily living activities was measured using Oswestry Disability Index (Ar-ODI).The questionnaire contains 10 items related to limitations in daily life activities (like personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and work).Each item includes six potential responses that are rating on a 0 to 5 points scale, with maximum scores of ''5'' or ''total disability'' and a minimum score of ''0'' or ''no disability.'' 39-41 The total score is calculated as follows: (patient' score/50) *100 to obtain the score expressed in percentage

OTHER OUTCOMES:
Assessment procedure of lumbar flexion and extension ROM | 4 weeks
  Two inclinometers were used to measure lumbar flexion and extension. The examiner stood behind the standing subject. The skin was marked along the spine midway between two posterior superior iliac spines (PSIS), and one mark was made on the spinous processes, 15 cm superior to the PSIS line. Both inclinometers were placed over the skin marks.

CONTACTS AND LOCATIONS:
Overall Officials: Rabab M Shoala, PHD, Principal Investigator — Basic Science Department, Faculty of Physical Therapy, Cairo University, Egypt.
Locations (1):
- Faculty of Physical Therapy, Cairo University., Cairo, Egypt, Egypt